CLINICAL TRIAL: NCT03307005
Title: Improving Sleep Quality in Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00142395
Record Dates: First submitted 2017-09-28; First posted 2017-10-11 (Actual); Results first posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Sleep Disturbance; Heart Failure
MeSH Terms: conditions — Parasomnias; Heart Failure | interventions — Zolpidem

STUDY DESIGN:
Intervention Model Description: Single-site, randomized, parallel, placebo controlled, double blind study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Drug: Zolpidem Tartrate
- Control (Placebo Comparator)
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Zolpidem Tartrate — Zolpidem tartrate 5 mg capsule one per night taken for 7 nights
  Arms: Intervention
Drug: Placebo oral capsule — Placebo capsule one per night taken for 7 nights
  Arms: Control

SUMMARY:
Poor sleep quality is common in patients with heart failure. The limited available evidence intimates that improving sleep quality in patients with heart failure may improve morbidity and quality of life in this patient population. However, there is a paucity of evidence assessing the use of effective pharmacologic therapies in heart failure. The nonbenzodiazepine, GABA receptor agonist, zolpidem, has been found to have considerable benefits over traditional benzodiazepines as a soporific medication. The investigators hypothesize that zolpidem will safely improve sleep quality in patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-79 years old
* HFrEF, EF ≤ 45% (by echocardiography)
* NYHA functional class I to III
* Able to give written consent
* On goal-directed medical therapy for HF, with stable dosing of HF medications for 2 weeks prior to enrollment
* No hospitalizations for HF within the past month
* Positive response to experiencing any of the following sleep-related symptoms at least once a week:
* Difficulty falling asleep
* Waking up during the night and having difficulty getting back to sleep
* Waking up too early in the morning and being unable to get back to sleep.

Exclusion Criteria:

* Use of sedative-hypnotics, anxiolytic, or benzodiazepines within the previous 2 weeks
* Current treatment with other sedating medications such as opioids
* On therapy for pharmacological therapy for depression
* History of alcohol/drug dependence
* History of liver disease, HIV, or severe COPD
* On Thorazine
* Current use of ketoconazole
* Current use of tricyclic antidepressants
* Current use of macrolide antibiotics
* Current use of anticonvulsant medications
* Pregnancy. A urine pregnancy test will be performed to exclude pregnancy in potential subjects.

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rashmi Aurora, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Campus, Asthma and Allergy Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo oral capsule: Placebo capsule one per night taken for 7 nights
Period: Overall Study
Arm/Group | Zolpidem Tartrate | Placebo
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Persons with heart failure and insomnia
Groups:
- Intervention: Participants received seven nights of zolpidem 5 mg
- Control: Participants received seven nights of placebo
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Continuous [Mean (Full Range); unit: years] | 60.3 [43 to 75] | 67.5 [65 to 70] | 63.2 [43 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 2 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Sleep Latency
Description: Mean change in sleep latency on second sleep study minus sleep latency on the first sleep study. Lower values suggest faster sleep onset. Sleep latency is measured in minutes.
Time Frame: 1 week
Measure: Mean (Full Range); unit: minutes
Arm/Group | Intervention | Control
Number analyzed (Participants) | 3 | 2
minutes | -73.3 [-143 to 0.2] | 21.9 [-5.5 to 49.1]

2. Primary Outcome: Total Sleep Time
Description: Mean change in total sleep time on second sleep study minus total sleep time on first sleep study. Higher values suggest more total sleep time. Total sleep time is measured in minutes.
Time Frame: 1 week
Measure: Mean (Full Range); unit: minutes
Arm/Group | Intervention | Control
Number analyzed (Participants) | 3 | 2
minutes | 67.8 [36.5 to 125.3] | -87.3 [-184.5 to 10]

3. Primary Outcome: Sleep Efficiency
Description: Mean change in sleep efficiency on second sleep study minus sleep efficiency on the first sleep study. Higher values suggest more efficient sleep. Sleep efficiency is described as a percentage.
Time Frame: 1 week
Measure: Mean (Full Range); unit: sleep efficiency percentage
Arm/Group | Intervention | Control
Number analyzed (Participants) | 3 | 2
sleep efficiency percentage | 7.3 [0 to 17] | -5.5 [-33 to 22]

4. Other Pre Specified Outcome: Insomnia Severity Index
Description: a questionnaire that assesses insomnia severity with a range of score from 0-28. Scores >=15 are signify the presence of insomnia
Time Frame: 1 week
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 3 | 2
score on a scale
  Baseline ISI score | 16.7 [11 to 24] | 14 [12 to 16]
  Final ISI score | 11 [4 to 23] | 13.5 [11 to 16]

5. Other Pre Specified Outcome: Kansas City Cardiomyopathy Questionnaire
Description: a validated, disease-specific quality of life measure for patients with heart failure. Raw scores vary from 22-133. Lower scores signify worst heart failure-related quality of life.
Time Frame: 1 week
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 3 | 2
score on a scale
  Baseline KCCQ-23 Score | 91.7 [77 to 120] | 99 [85 to 113]
  Final KCCQ-23 Score | 97.3 [80 to 117] | 100 [95 to 105]

6. Other Pre Specified Outcome: Epworth Sleepiness Scale
Description: a validated questionnaire that assesses chronic subjective sleepiness. The scale ranges from 0-24 with higher values signifying more sleepiness. A binary cutpoint of 11 or higher is considered significant sleepiness.
Time Frame: 1 week
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 3 | 2
score on a scale
  Baseline ESS score | 10.3 [5 to 16] | 12.5 [8 to 17]
  Final ESS score | 7 [1 to 16] | 13 [7 to 19]

7. Other Pre Specified Outcome: Pittsburgh Sleep Quality Index
Description: a self report questionnaire that assess sleep quality. The scale ranges from 0-21. Scores higher than 5 indicate poor sleep quality
Time Frame: 1 week
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 3 | 2
score on a scale
  Baseline PSQI score | 10.7 [8 to 14] | 12 [10 to 14]
  Final PSQI score | 11.3 [9 to 15] | 11 [10 to 12]

ADVERSE EVENTS:
Time Frame: 15 months.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/05/NCT03307005/Prot_SAP_001.pdf